CLINICAL TRIAL: NCT03084185
Title: Evaluation of the Role of Plasma Biomarkers for Portal Hypertension Progression and Oxidative Damage in Decompensation of Cirrhotic Patient.
Brief Title: Evaluation of the Role of Plasma Biomarkers in the Development of Decompensation in Patients With Cirrhosis .
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, ERICA VILLA, Professor, University of Modena and Reggio Emilia
Other Study IDs: HVPG_HCV
Record Dates: First submitted 2017-03-08; First posted 2017-03-20 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-03

CONDITIONS: Cirrhosis
Keywords: decompensation; deficit; metabolomics; portal hypertension
MeSH Terms: conditions — Fibrosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-center and prospective study to identify specific biomarker in order to predict development of decompensation in cirrhotic patients.

The duration of the study is 36 months and it provides a cohort of 200 patients.

DETAILED DESCRIPTION:
At screening, patient will have taken blood samples and performed hepatic vein pressure gradient.

After randomization, patient will be seen at follow up every 3 months to do blood sample and every 12 months to undergo hepatic vein pressure gradient , according to the guidelines.

In addition, metabolomics analysis will be performed at screening and every 3 months. The results will be analyzed in relation to emergence of decompensation during follow up period, in order to identify specific metabolomics characteristics that may be able to predict decompensation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of liver cirrhosis
* Aged between 18 and 75 years
* Obtaining written informed consent
* Absence of exclusion criteria

Exclusion Criteria:

* Diagnosis of hepatocellular carcinoma
* Presence of portal vein thrombosis
* HIV
* Liver transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with cirrhosis
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Identification of predictive biomarkers for the deficit development in patients with compensated cirrhosis. | December 2018
  Patients will be subject to blood sample periodically and following exams will be made:
  * Chemistry and hematology to define liver function
  * Intestinal Fatty Acid Binding Protein
  * 16S, ribosomal deoxyribonucleic acid
  * Cluster of differentiation 14
  * Interleukin 6
  * Asymmetrical dimethylarginine
  * Tissue factor
  According to current guidelines, patients will be submitted to:
  * Hepatic vein pressure gradient AND combined right heart catheterization
  * Liver elastography

SECONDARY OUTCOMES:
Finding of serum metabolomic features of cirrhotic patients. | December 2018
  Analysis will be conducted on sera collected during the screening and every three months. These samples will be examined using liquid chromatography and mass spectrometry in order to obtain the identification of main components and their mass than, the informations will be analyzed by MarkerLynxTM software

CONTACTS AND LOCATIONS:
Overall Officials: ERICA VILLA, MD, Principal Investigator — University of Modena and Reggio Emilia
Locations (1):
- Azienda Ospedaliera Universitaria Policlinico Di Modena, Modena, MO, Italy

IPD SHARING:
Plan to Share IPD: No